CLINICAL TRIAL: NCT07295509
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II/III Clinical Study to Evaluate the Efficacy and Safety of Picankibart in Patients With Active Psoriatic Arthritis
Brief Title: A Study of Picankibart in Patients With Active Psoriatic Arthritis
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Innovent Biopharmaceutical Technology (Hangzhou) Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI112C301
Record Dates: First submitted 2025-11-24; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Picankibart Group 2 (Experimental): Participants receive picankibart SC at each scheduled dosing timepoint with dosing interval 2.
  Interventions: Other: Placebo; Drug: Picankibart
- Placebo Group (Placebo Comparator): Participants receive placebo SC at each scheduled dosing timepoint. Treatment of picankibart starts at Week 26.
  Interventions: Other: Placebo; Drug: Picankibart
- Picankibart Group 1 (Experimental): Participants receive picankibart SC at each scheduled dosing timepoint with dosing interval 1.
  Interventions: Drug: Picankibart

INTERVENTIONS:
Other: Placebo — Placebo administered SC at each scheduled dosing timepoint.
  Arms: Picankibart Group 2; Placebo Group
Drug: Picankibart — Picankibart administered SC at each scheduled dosing timepoint.

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase II/III clinical trial evaluating the efficacy and safety of picankibart (IBI112) in patients with active psoriatic arthritis (PsA). The study consists of two stages: Phase II dose-finding (n=90) and Phase III confirmatory (n=132). Participants will receive subcutaneous (SC) injections of either picankibart (200mg) or placebo with different dosing schedules, with placebo crossover to active treatment at Week 26. The Phase II portion will identify optimal dosing for Phase III, which will confirm efficacy. The study will evaluate improvements in joint symptoms, physical function, quality of life, and skin manifestations. Primary endpoint is percentage of participants who achieved an American College of Rheumatology (ACR) 20 Response at Week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Diagnosed with PsA for ≥6 months, and meeting Classification Criteria for Psoriatic Arthritis (CASPAR) at screening
3. Having active PsA: ≥3 tender joints and ≥3 swollen joints at screening and baseline, with CRP ≥3 mg/L at screening
4. Having active plaque psoriasis (≥1 lesion ≥2cm) or nail psoriasis, or a documented history of plaque psoriasis
5. Inadequate response or intolerance to prior NSAIDs or non-biologic DMARDs
6. Prior use of TNF-α inhibitors, IL-17/23 inhibitors, or JAK inhibitors is permitted if subjects exhibited inadequate response or intolerance, with an appropriate washout period
7. Stable doses of protocol permitted background therapy (if any)

Exclusion Criteria:

1. Other inflammatory conditions that may affect the evaluation of the study drug
2. Prior treatment with >2 biologic agents
3. Recent use of prohibited medications (specific washout periods apply)
4. Non-plaque psoriasis forms or drug-induced psoriasis
5. Severe, progressive, or uncontrolled renal, hepatic, cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, hematological, rheumatic (excluding PsA), psychiatric, or genitourinary conditions
6. Significant laboratory abnormalities
7. Pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who achieved an American College of Rheumatology (ACR) 20 response | Week 26
  The ACR20 response is defined as ≥20% improvement in swollen joint count (66 joints) and tender joint count (68 joints) and ≥20% improvement in 3 of following 5 assessments: participant's assessment of pain using Visual Analog Scale (VAS; 0-100 millimeter [mm], 0 mm=no pain and 100 mm=worst possible pain), participant's global assessment of disease activity by using VAS (scale ranges from 0 mm to 100 mm, [0 mm= very well to 100 mm= very poor]), physician's global assessment of disease activity using VAS (scale ranges from 0 to 100), [0 = no arthritis to 100 = extremely active arthritis], participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and C-reactive protein (CRP).

SECONDARY OUTCOMES:
Change from baseline in Disease Activity Score in 28 Joints (DAS28)-CRP score | Week 26, and from baseline to Week 56
  The DAS28-CRP is a measure of disease activity based on swollen and tender joint counts in 28 joints, CRP and the participant's global assessment of disease activity. The range of DAS28-CRP score is 0-10. Higher score means more disease activity.
Percentage of participants who achieved an ACR50 response | Week 26, and from baseline to Week 56
  The ACR50 response is defined as ≥50% improvement in swollen joint count (66 joints) and tender joint count (68 joints) and ≥50% improvement in 3 of following 5 assessments: participant's assessment of pain using Visual Analog Scale (VAS; 0-100 millimeter [mm], 0 mm=no pain and 100 mm=worst possible pain), participant's global assessment of disease activity by using VAS (scale ranges from 0 mm to 100 mm, [0 mm= very well to 100 mm= very poor]), physician's global assessment of disease activity using VAS (scale ranges from 0 to 100), [0 = no arthritis to 100 = extremely active arthritis], participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and C-reactive protein (CRP).
Percentage of participants who achieved an ACR70 response | Week 26, and from baseline to Week 56
  The ACR70 response is defined as ≥70% improvement in swollen joint count (66 joints) and tender joint count (68 joints) and ≥70% improvement in 3 of following 5 assessments: participant's assessment of pain using Visual Analog Scale (VAS; 0-100 millimeter [mm], 0 mm=no pain and 100 mm=worst possible pain), participant's global assessment of disease activity by using VAS (scale ranges from 0 mm to 100 mm, [0 mm= very well to 100 mm= very poor]), physician's global assessment of disease activity using VAS (scale ranges from 0 to 100), [0 = no arthritis to 100 = extremely active arthritis], participant's assessment of physical function measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area) and C-reactive protein (CRP).
Change from baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) | Week 26, and from baseline to Week 56
  HAQ-DI measures improvement in physical function/disability. It is defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area.
Change from baseline in Short Form Health Survey 36 (SF-36) Physical Component Summary (PCS) score | Week 26, and from baseline to Week 56
  The SF-36 Health determined participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 comprise the physical component of the SF-36. Scores on each item were summed and averaged (range = 0-100) and a positive change from Baseline indicates improvement.
Enthesitis/dactylitis resolution rates | Week 26, and from baseline to Week 56
  Percentage of participants with complete resolution of enthesitis (inflammation at tendon/ligament attachments) or dactylitis (sausage-digit swelling).
Percentage of participants who achieved 75%Psoriasis Area and Severity Index 75 response | From baseline to Week 56
  Percentage of participants who achieve at least 75% or 90% or 100% reduction in Psoriasis Area and Severity Index (PASI) score, assessing skin lesion severity in psoriatic arthritis patients.
Change from baseline in van der Heijde-modified Total Sharp Score (vdH-mTSS) | Week 26 and Week 56
  The vdH-mTSS is a measure of change in joint health. X-rays of hands and feet are obtained at screening, Week 26 and Week 56. Totals for hands and feet for erosion scores (range 0 to 320) and joint space narrowing scores (range 0 to 208) were calculated and added to obtain the vdH-mTSS (range = 0 [normal] to 528 [maximal disease]). An increase in vdH-mTSS from baseline represents disease progression and/or joint worsening.
Percentage of participants who experienced adverse events (AEs) | From baseline to Week 56
  An AE is any untoward medical occurrence, which does not necessarily have a causal relationship with treatment.
Percentage of participants who experienced serious adverse events (SAEs) | From baseline to Week 56
  An SAE is an AE that results in death, is life-threatening, results in or prolongs hospitalization, results in congenital anomaly, persistent or significant disability/incapacity, spontaneous or elective abortion, or requires intervention to prevent a serious outcome.
Maximum plasma concentration (Cmax) of picankibart | From baseline to Week 56
  Plasma concentration of picankibart is evaluated at each scheduled dosing timepoint. Cmax is the highest concentration of a drug in the blood.
Area under the concentration-time curve (AUC) of picankibart | From baseline to Week 56
  Plasma concentration of picankibart is evaluated at each scheduled dosing timepoint. AUC represents the area under the concentration-time curve and gives insight into the extent of exposure to a drug and its clearance rate from the body.
Percentage of participants who developed anti-drug antibody (ADA) | From baseline to Week 56
  ADAs are immune system-produced antibodies that specifically bind to therapeutic drugs, potentially altering their pharmacokinetics, efficacy, or safety.
Percentage of participants who developed neutralizing antibody (NAb) | From baseline to Week 56
  NAbs are ADAs that inhibit the drug's biological function by blocking target interaction.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China